CLINICAL TRIAL: NCT02774031
Title: Comparing Gas Consumption With Conventional Low Flow Ventilation and Gas Control Systems From Two Different Anesthesia Machines: Flow-i and Aisys
Brief Title: Comparison of Gas Consumption From Two Different Anesthesia Machines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/2132
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Male Urogenital Diseases; Female Urogenital Diseases
Keywords: Anesthesia, Inhalation; Laparoscopy; Prostatectomy; Cystectomy; Gynecologic Surgical Procedures
MeSH Terms: conditions — Male Urogenital Diseases; Female Urogenital Diseases; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aisys with Et control (Experimental): the ventilation modus will be pressure control ventilation with volume guarantee (PCV-VG). Settings: tidal volume (TV) 7-9 ml/kg BW, respiratory rate (RR) 12 -14/min, and 8-10 cmH2O positive end expiratory pressure (PEEP). Target for end expired desflurane concentration (F A des) is set to 4.2%, and target for end expired oxygen (F AO2) is set to 35%.
  Interventions: Device: Aisys with Et control
- Aisys conventional ventilation (Active Comparator): 50% oxygen and 50% air in 1 liter FGF will be administered. To be started with a FGF of 5l/min and vaporizer setting at 6 Vol% for 5 min. Then the FGF will be reduced to 1 l/min. 25 min later the vaporizer setting will be reduced to 5.5 Vol % for the rest of the study period. Ventilation modus for this group will be the same as for 'Aisys with PCV-VG'
  Interventions: Device: Aisys conventional
- Flow-i with ACG (Experimental): the following parameters will be preset: FIO2= 40%; end expired gas concentration (FA des) to 4.2%; speed 6; and ventilation modus = pressure regulated volume control (PRVC) with tidal volume (TV) 7-9 ml/kg BW, respiratory rate (RR)12-14/min, and 8-10 cmH2O positive end expiratory pressure (PEEP).
  Interventions: Device: Flow-i with ACG
- Flow-I conventional ventilation (Active Comparator): 50% oxygen and 50% air in 1 liter FGF will be administered. To be started with a FGF of 5l/min and vaporizer setting at 6 Vol% for 5 min. Then the FGF will be reduced to 1 l/min. 25 min later the vaporizer setting will be reduced to 5.5 Vol % for the rest of the study period. Ventilation modus for this group will be the same as for 'Flow-i with ACG'
  Interventions: Device: Flow-i conventional

INTERVENTIONS:
Device: Aisys with Et control
  Arms: Aisys with Et control
Device: Aisys conventional
  Arms: Aisys conventional ventilation
Device: Flow-i with ACG
  Arms: Flow-i with ACG
Device: Flow-i conventional
  Arms: Flow-I conventional ventilation

SUMMARY:
Low flow anesthesia (LFA) is used less than desirable, partly because one has considered that there might be danger of underdosing of anesthesia gas and thus risk of awareness under anesthesia.LFA has several advantages such as reducing loss of moisture and heat in the inhaled air under anesthesia and to reduce the consumption of anesthetic gas. A few anesthesia machines include an automatic gas control system: the Aisys machine, by GE Healthcare (Madison, WI, USA), and the Flow-i machine, by Maquet (Sweden).

Since these machines were introduced, only a few studies have reported their functionality and effect on gas consumption. 20 to 55% reduction of gas consumption was found. The potential reduction may have been underestimated because in the majority of cases a FGF higher than 1 l/min was still used.

In this study the consumption of anesthetic gas (desflurane) delivered by two different anesthesia machines (Aisys and Flow-i) will be compared, with and without gas control delivery systems. Gas consumption and the time needed to reach the target level of anesthetic gas concentration will be assessed. Data needed will be collected directly from the anesthesia machine, PICIS ( Electronic anesthesia record) and EPJ (Electronic patient journal). The results of this study are of interest for intraoperative ventilation and of economic and ecological interest

.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robot assisted laparoscopic prostatectomy, robot assisted laparoscopic cystectomy or robot assisted laparoscopic gynecological surgery

Exclusion Criteria:

* Cognitive failure, which compromises the ability for an informed consent.
* Pregnancy
* American Society of Anesthesiologists physical status classification system (ASA) IV-VI

Patients who are included in the study can be excluded for the following reasons:

* surgical technical problems (for example surgically impossible to complete the operation with robot assisted surgery)
* technical problems with the anesthesia machine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
gas consumption in ml/hr | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Pål Klepstad, PhD MD, Study Director — St. Olavs Hospital
Locations (1):
- Department of Anesthesia, St.Olavs University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided